CLINICAL TRIAL: NCT04278248
Title: A Randomized, Blinded, Parallel Controlled, Phase Ⅲ Clinical Trial to Evaluate Immunogenicity and Safety of 23-Valent Pneumococcal Polysaccharide Vaccine in Healthy Volunteers Aged 2 Years and Above
Brief Title: Immunogenicity and Safety of 23-Valent Pneumococcal Polysaccharide Vaccine in Healthy Volunteers Aged 2 Years and Above
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201719906
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Received Vaccine: 23-valent Pneumococcal Polysaccharide Vaccine(experimental vaccine), 0.5 ml/dose
  Interventions: Biological: 23-Valent Pneumococcal Polysaccharide Vaccine
- Positive control group (Active Comparator): Received Vaccine: 23-valent Pneumococcal Polysaccharide Vaccine (positive control vaccine), 0.5 ml/dose
  Interventions: Biological: 23-Valent Pneumococcal Polysaccharide Vaccine

INTERVENTIONS:
Biological: 23-Valent Pneumococcal Polysaccharide Vaccine — 1 dose according to age of subjects. Single intramuscular dose contains 0.5ml 23-Valent Pneumococcal Polysaccharide Vaccine.

SUMMARY:
The purpose of this study is to evaluate Immunogenicity and safety of 23-Valent Pneumococcal Polysaccharide Vaccine in healthy volunteers aged 2 Years and above.

ELIGIBILITY:
Inclusion Criteria:

* 2 years old and above healthy people.
* Subject or legal representative who consent and has signed written informed consent.
* Subject or legal representative who is able to comply with all study procedures.
* Subject who didn't vaccinate pneumococcal vaccines and did't immune with any live vaccine within 14 days and inactivated vaccine within 7 days before vaccination.
* Axillary temperature ≤37.0 ℃.

Exclusion Criteria:

* History of allergy，eclampsia, epilepsy, encephalopathy and mental disease or family disease.
* Allergic history after vaccination.
* Known allergy to any component of the test vaccine（the test vaccine mainly contains 23 types of pneumococcal polysaccharide and PBS buffer）
* Subjects who diagnosis of thrombocytopenia or other history of coagulopathy.
* Known immunological impairment or dysfunction.
* Subjects who have received whole blood, plasma, and immunoglobulin therapy within one month.
* Known severe congenital malformations, developmental disorders; clinically diagnosed serious chronic diseases: down's syndrome, diabetes, sickle cell anemia or neurological disorders, Guillain Barre syndrome.
* Known or suspected to suffer from: respiratory system disease，acute infection or chronic disease active period，severe cardiovascular disease, liver and kidney disease, malignant tumor, skin disease,children's mother has HIV infection and other serious and infectious diseases.
* In pregnancy or lactation or pregnant women.
* Subjects aged 18 years and above whose systolic blood pressure≥160mmHg and diastolic blood pressure≥100mmHg.
* Any contraindications that investigators consider related to vaccination.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1940 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity study endpoint | 30 day after each vaccination
  Percentage of participants with seroresponse to each vaccination
Safety study endpoint | 30 day after each vaccination
  Occurrence of adverse events during a 30 day follow-up period after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Du Lin, Master, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Yizhou Center for Disease Control and Prevention, Yizhou, Guangxi, China

IPD SHARING:
Plan to Share IPD: No